CLINICAL TRIAL: NCT01932606
Title: Acute Effects of Inorganic Nitrite on Cardiovascular Hemodynamics in Heart Failure With Preserved Ejection Fraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barry Borlaug (Other)
Responsible Party: Sponsor-Investigator, Barry Borlaug, M.D., Associate Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-004077
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Heart Disease; Heart Failure With Preserved Ejection Fraction; Exercise Intolerance; Pulmonary Hypertension
MeSH Terms: conditions — Heart Diseases; Hypertension, Pulmonary | interventions — Nitrites

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrite (Experimental): Study drug (NaNO_2 50 mcg/kg/min) will be infused for 5 minutes during the cardiac catheterization procedure.
  Interventions: Drug: Nitrite
- Saline (Placebo Comparator): Saline Placebo for Nitrite will be infused for 5 minutes during the cardiac catheterization procedure.
  Interventions: Drug: Saline Placebo for Nitrite

INTERVENTIONS:
Drug: Nitrite — Study drug (NaNO_2 50 mcg/kg/min) will be infused for 5 minutes during the cardiac catheterization procedure.
  Arms: Nitrite
Drug: Saline Placebo for Nitrite — Normal saline placebo will be infused for 5 minutes during the cardiac catheterization procedure. Hemodynamics will then be measured at baseline after study drug infusion and again during low level exercise (20 Watts).
  Arms: Saline

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is a major public health problem that has no proven effective treatment. This study assessed the effects of acute nitrite administration on resting and exercise hemodynamics in patients with HFpEF.

DETAILED DESCRIPTION:
Subjects were studied on their long-term medications in the post-absorptive state and supine position. Right heart catheterization was performed with simultaneous expired gas analysis at rest and during supine exercise at a 20 Watts workload for 5 minutes. After the first exercise phase (before any drug administration) and after return to steady-state baseline hemodynamic values, subjects were randomized. Study drug or placebo was infused for 5 minutes. After a 10 minute observation period, hemodynamic measurements were repeated at rest, followed by repeat supine exercise at a 20 Watts workload for 5 minutes, identical to the study's first phase. Arterial and venous blood samples and hemodynamic and expired gas data were acquired during each stage of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a cardiac catheterization procedure.
* Clinical symptoms of shortness of breath and fatigue
* Normal left ventricular ejection fraction (≥50%)
* Elevated left ventricular filling pressures at cardiac catheterization (defined as resting pulmonary capillary wedge pressure (PCWP)>15 mmHg and/or PCWP≥25 mmHg during exercise)

Exclusion Criteria:

* Systolic BP <120 mmHg
* Prior nitrate therapy (within previous 2 weeks)
* Glucose 6-phosphate dehydrogenase (G6PD) deficiency
* Other "non-HFpEF" specific causes of heart failure such as significant valvular disease (>moderate left-sided regurgitation, >mild stenosis), severe pulmonary disease, unstable coronary disease or coronary spasm, primary renal or hepatic disease, constrictive pericarditis, or infiltrative, restrictive, or hypertrophic cardiomyopathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Borlaug BA, Koepp KE, Melenovsky V. Sodium Nitrite Improves Exercise Hemodynamics and Ventricular Performance in Heart Failure With Preserved Ejection Fraction. J Am Coll Cardiol. 2015 Oct 13;66(15):1672-82. doi: 10.1016/j.jacc.2015.07.067. PMID 26449137
- [Derived] Reddy YNV, Stewart GM, Obokata M, Koepp KE, Borlaug BA. Peripheral and pulmonary effects of inorganic nitrite during exercise in heart failure with preserved ejection fraction. Eur J Heart Fail. 2021 May;23(5):814-823. doi: 10.1002/ejhf.2093. Epub 2021 Feb 1. PMID 33421267

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in the trial between January and September 2014.
Groups:
- Placebo: Saline Placebo for Nitrite will be infused for 5 minutes during the cardiac catheterization procedure.
Period: Overall Study
Arm/Group | Nitrite | Placebo
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitrite | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (6) | 70 (8) | 69 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Exercise Pulmonary Capillary Wedge Pressure (PCWP)
Description: Pulmonary capillary wedge pressure (PCWP) provides an indirect estimate of left atrial pressure (LAP). PCWP is the pressure measured by wedging a pulmonary catheter with an inflated balloon into a small pulmonary arterial branch.
Time Frame: during repeat exercise run, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
mm Hg | 19.0 (5.0) | 28.0 (6.0)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Test type: Superiority or Other; p = 0.0003, ANCOVA

2. Secondary Outcome: Change in Central Pressures After Study Drug (Resting)
Description: Values are resting values after receiving study drug minus resting values before study drug (on the same day.)
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
mm Hg
  Right atrial pressure | -2 (2) | 0 (1)
  Pulmonary artery systolic pressure | -8 (5) | -3 (4)
  Mean pulmonary artery pressure | -6 (3) | -1 (3)
  PCWP | -3 (3) | 0 (1)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in right atrial pressure; Test type: Superiority or Other; p = 0.0003, t-test, 2 sided
Statistical Analysis 2: Comparison: Nitrite vs Placebo; Comparison between the arms for change in pulmonary artery systolic pressure; Test type: Superiority or Other; p = 0.01, t-test, 2 sided
Statistical Analysis 3: Comparison: Nitrite vs Placebo; Comparison between the arms for change in mean pulmonary artery pressure; Test type: Superiority or Other; p = 0.002, t-test, 2 sided
Statistical Analysis 4: Comparison: Nitrite vs Placebo; Comparison between the 2 arms for change in PCWP; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Change in Heart Rate After Study Drug (Resting)
Description: Values are resting values after receiving study drug minus resting values before study drug (on the same day.)
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
beats/minute | 0 (5) | -3 (5)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Test type: Superiority or Other; p = 0.15, t-test, 2 sided

4. Secondary Outcome: Change in Blood Pressure After Study Drug (Resting)
Description: Values are resting values after receiving study drug minus resting values before study drug (on the same day.)
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
mm Hg
  Systolic Blood Pressure | -7 (8) | -2 (10)
  Mean Blood Pressure | -3 (4) | -1 (6)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in systolic blood pressure; Test type: Superiority or Other; p = 0.11, t-test, 2 sided
Statistical Analysis 2: Comparison: Nitrite vs Placebo; Comparison between the arms for change in mean blood pressure; Test type: Superiority or Other; p = 0.2, t-test, 2 sided

5. Secondary Outcome: Change in Pulmonary Vascular Resistance (PVR) After Study Drug (Resting)
Description: Values are resting values after receiving study drug minus resting values before study drug (on the same day.) Pulmonary Vascular Resistance (PVR) is the resistance to flow that must be overcome to push blood through the pulmonary vasculature. Acute and chronic lung disease can both cause an increase in PVR. Chronic PVR can lead to right sided heart failure.
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: mm Hg/L/min
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
mm Hg/L/min | -0.3 (0.4) | -0.4 (0.6)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in PVR; Test type: Superiority or Other; p = 0.7, t-test, 2 sided

6. Secondary Outcome: Change in Pulmonary Artery (PA) Compliance After Study Drug (Resting)
Description: Values are resting values after receiving study drug minus resting values before study drug (on the same day.) Pulmonary artery compliance is an index of the elasticity of the blood vessel, an indication of arterial stiffness.
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: ml/mm Hg
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
ml/mm Hg | 0.8 (1.3) | 0.2 (0.6)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in pulmonary artery compliance; Test type: Superiority or Other; p = 0.1, t-test, 2 sided

7. Secondary Outcome: Change in Systemic Vascular Resistance (SVR) After Study Drug (Resting)
Description: Values are resting values after receiving study drug minus resting values before study drug (on the same day.) Systemic vascular resistance (SVR) refers to the resistance to blood flow offered by all of the systemic vasculature, excluding the pulmonary vasculature.
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: dyne/s * cm^5
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
dyne/s * cm^5 | 140 (350) | 20 (160)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in SVR; Test type: Superiority or Other; p = 0.3, t-test, 2 sided

8. Secondary Outcome: Change in Left Ventricular Stroke Work (LVSW) After Study Drug (Resting)
Description: Values are resting values after receiving study drug minus resting values before study drug (on the same day.) Stroke work refers to the work done by the ventricle to eject a volume of blood (i.e., stroke volume) into the aorta. Ventricular stroke work can be estimated as the product of stroke volume and mean aortic pressure during ejection.
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: g/beat
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
g/beat | -6 (18) | 0 (9)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in LVSW; Test type: Superiority or Other; p = 0.3, t-test, 2 sided

9. Secondary Outcome: Change in Oxygen Consumption (VO_2) After Study Drug (Resting)
Description: Values are resting values after receiving study drug minus resting values before study drug (on the same day.)
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
ml/min | -2 (38) | -6 (15)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in VO_2; Test type: Superiority or Other; p = 0.8, t-test, 2 sided

10. Secondary Outcome: Change in Arteriovenous Oxygen Content Difference After Study Drug (Resting)
Description: Values are resting values after receiving study drug minus resting values before study drug (on the same day.) Arteriovenous oxygen difference is the difference in the oxygen content of the blood between the arterial blood and the venous blood. It is an indication of how much oxygen is removed from the blood in capillaries as the blood circulates in the body.
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: ml/dl
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
ml/dl | 0.4 (0.5) | 0 (0.4)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for arteriovenous oxygen content difference; Test type: Superiority or Other; p = 0.1, t-test, 2 sided

11. Secondary Outcome: Change in Cardiac Output After Study Drug (Resting)
Description: Values are resting values after receiving study drug minus resting values before study drug (on the same day.) The volume of blood pumped per minute by each ventricle of the heart. Cardiac output is equal to the stroke volume (the amount of blood pumped from a ventricle in a single heartbeat) times the heart rate.
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
L/min | -0.4 (0.8) | -0.2 (0.5)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in cardiac output; Test type: Superiority or Other; p = 0.4, t-test, 2 sided

12. Secondary Outcome: Change in Stroke Volume After Study Drug (Resting)
Description: Values are resting values after receiving study drug minus resting values before study drug (on the same day.) Stroke volume is the amount of blood pumped out of the heart (left ventricle - to the body) during each contraction.
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
ml | -5 (16) | -1 (9)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in stroke volume; Test type: Superiority or Other; p = 0.4, t-test, 2 sided

13. Secondary Outcome: Change in Central Pressures After Study Drug (Exercise)
Description: Values are exercise values after receiving study drug minus exercise values before study drug (on the same day.)
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
mm Hg
  Right atrial pressure | -5 (2) | -1 (2)
  Pulmonary artery systolic pressure | -11 (6) | -4 (8)
  Mean pulmonary artery pressure | 10 (4) | -2 (5)
  PCWP | -11 (5) | -2 (5)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in right atrial pressure (exercise); Test type: Superiority or Other; p = 0.0002, t-test, 2 sided
Statistical Analysis 2: Comparison: Nitrite vs Placebo; Comparison between the arms for change in pulmonary artery systolic pressure (exercise); Test type: Superiority or Other; p = 0.01, t-test, 2 sided
Statistical Analysis 3: Comparison: Nitrite vs Placebo; Comparison between the arms for change in mean pulmonary artery pressure (exercise); Test type: Superiority or Other; p = 0.0002, t-test, 2 sided
Statistical Analysis 4: Comparison: Nitrite vs Placebo; Comparison between the arms for change in PCWP (exercise); Test type: Superiority or Other; p = 0.0002, t-test, 2 sided

14. Secondary Outcome: Change in Heart Rate After Study Drug (Exercise)
Description: Values are exercise values after receiving study drug minus exercise values before study drug (on the same day.)
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
beats/minute | -1 (6) | 0 (3)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in heart rate; Test type: Superiority or Other; p = 0.3, t-test, 2 sided

15. Secondary Outcome: Change in Blood Pressure After Study Drug (Exercise)
Description: Values are exercise values after receiving study drug minus exercise values before study drug (on the same day.)
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
mm Hg
  Systolic Blood Pressure | -5 (13) | 2 (10)
  Diastolic Blood Pressure | -5 (8) | 0 (2)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in systolic blood pressure; Test type: Superiority or Other; p = 0.2, t-test, 2 sided
Statistical Analysis 2: Comparison: Nitrite vs Placebo; Comparison between the arms for change in diastolic blood pressure; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

16. Secondary Outcome: Change in PVR After Study Drug (Exercise)
Description: Values are exercise values after receiving study drug minus exercise values before study drug (on the same day.) Pulmonary Vascular Resistance (PVR) is the resistance to flow that must be overcome to push blood through the pulmonary vasculature. Acute and chronic lung disease can both cause an increase in PVR. Chronic PVR can lead to right sided heart failure.
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: mm Hg/L/min
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
mm Hg/L/min | 0 (0.4) | 0.2 (0.4)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in PVR after study drug (exercise); Test type: Superiority or Other; p = 0.3, t-test, 2 sided

17. Secondary Outcome: Change in PA Compliance After Study Drug (Exercise)
Description: Values are exercise values after receiving study drug minus exercise values before study drug (on the same day.) Pulmonary artery compliance is an index of the elasticity of the blood vessel, an indication of arterial stiffness.
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: ml/mm Hg
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
ml/mm Hg | 0.8 (0.9) | 0.5 (0.9)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in PA compliance after study drug (exercise); Test type: Superiority or Other; p = 0.3, t-test, 2 sided

18. Secondary Outcome: Change in SVR After Study Drug (Exercise)
Description: Values are exercise values after receiving study drug minus exercise values before study drug (on the same day.) Systemic vascular resistance (SVR) refers to the resistance to blood flow offered by all of the systemic vasculature, excluding the pulmonary vasculature.
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: dyne/s * cm^5
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
dyne/s * cm^5 | -70 (140) | 70 (100)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in SVR after study drug (exercise); Test type: Superiority or Other; p = 0.007, t-test, 2 sided

19. Secondary Outcome: Change in LVSW After Study Drug (Exercise)
Description: Values are exercise values after receiving study drug minus exercise values before study drug (on the same day.) Stroke work refers to the work done by the ventricle to eject a volume of blood (i.e., stroke volume) into the aorta. Ventricular stroke work can be estimated as the product of stroke volume and mean aortic pressure during ejection.
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: g/beat
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
g/beat | 15 (12) | -2 (8)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in LVSW after study drug (exercise); Test type: Superiority or Other; p = 0.0003, t-test, 2 sided

20. Secondary Outcome: Change in Oxygen Consumption (VO_2) After Study Drug (Exercise)
Description: Values are exercise values after receiving study drug minus exercise values before study drug (on the same day.)
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
ml/min | 70 (138) | -30 (67)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in oxygen consumption (VO_2) after study drug (exercise); Test type: Superiority or Other; p = 0.02, t-test, 2 sided

21. Secondary Outcome: Change in Arteriovenous Oxygen Difference After Study Drug (Exercise)
Description: Arteriovenous oxygen difference is the difference in the oxygen content of the blood between the arterial blood and the venous blood. It is an indication of how much oxygen is removed from the blood in capillaries as the blood circulates in the body.
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: ml/dl
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
ml/dl | 0.2 (0.4) | 0 (0.6)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in arteriovenous oxygen difference after study drug (exercise); Test type: Superiority or Other; p = 0.6, t-test, 2 sided

22. Secondary Outcome: Change in Cardiac Output After Study Drug (Exercise)
Description: Values are exercise values after receiving study drug minus exercise values before study drug (on the same day.) Cardiac output is equal to the stroke volume (the amount of blood pumped from a ventricle in a single heartbeat) times the heart rate.
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
L/min | 0.5 (0.7) | -0.4 (0.7)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in cardiac output after study drug (exercise); Test type: Superiority or Other; p = 0.002, t-test, 2 sided

23. Secondary Outcome: Change in Stroke Volume After Study Drug (Exercise)
Description: Values are exercise values after receiving study drug minus exercise values before study drug (on the same day.) Stroke volume is the amount of blood pumped out of the heart (left ventricle - to the body) during each contraction.
Time Frame: baseline, approximately 30 minutes after study drug administration
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 14 | 14
ml | 7 (8) | -5 (6)
Statistical Analysis 1: Comparison: Nitrite vs Placebo; Comparison between the arms for change in stroke volume after study drug (exercise); Test type: Superiority or Other; p = 0.0002, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Subjects will be followed for adverse event reporting during the procedure and the recovery period, approximately 3 hours after the procedure on Day 1.
Arm/Group | Nitrite | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes